CLINICAL TRIAL: NCT01483924
Title: A 12-week Randomized, Double-blind, Placebo-controlled, Multicenter, Multiple Sequential Dose Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Apo805K1 in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Study to Evaluate Apo805K1 in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP03-0210
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Plaque Psoriasis
Keywords: Mild to Moderate Chronic Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 10 mg Apo805K1, or placebo (Experimental)
  Interventions: Drug: Apo805K1
- 30 mg Apo805K1, or placebo (Experimental)
  Interventions: Drug: Apo805K1
- 60 mg Apo805K1, or placebo (Experimental)
  Interventions: Drug: Apo805K1
- 100 mg Apo805K1, or placebo (Experimental)
  Interventions: Drug: Apo805K1

INTERVENTIONS:
Drug: Apo805K1 — Sequential parallel dose escalation.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of 12 weeks of treatment with Apo805K1 in subjects with moderate to severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
A) To evaluate the safety and tolerability of 12 weeks of treatment with Apo805K1

B) To evaluate the pharmacokinetics of Apo805K1 following daily administration for 14 days

C) To evaluate the efficacy and pharmacodynamics of Apo805K1

ELIGIBILITY:
Main Inclusion Criteria:

* A clinical diagnosis of moderate to severe chronic plaque psoriasis for at least 6 months (before Baseline assessment) with current body surface area (BSA) involvement ≥10% and Psoriasis Area Severity Index (PASI) ≥10.
* Male and female subjects 18 to 65 years of age, inclusive.
* At least one psoriatic plaque ≥6 mm in diameter (in a location suitable for biopsy).
* Signed and witnessed written informed consent form obtained prior to the first study intervention, as well as the ability to adhere to study restrictions, appointments and evaluation schedule.

Main Exclusion Criteria:

* Treatment of psoriasis with biologic agents within 90 days prior to Baseline assessment and during the study.
* Treatment with methotrexate, cyclosporine, retinoids, hydroxyurea or other systemic agents within 30 days prior to Baseline assessment and during the study.
* Phototherapy within 30 days prior to Baseline assessment and during the study.
* Psoriasis topical therapy within 14 days prior to Baseline assessment and during the study (exception: non-medicated emollients and tar shampoo will be allowed).
* History of liver disease or abnormal liver enzymes
* Serum creatinine ≥1.5 times the upper limit of normal for age and sex-matched controls.
* Previous treatment with Apo805K1or Thymodepressin or other immunosuppressant drugs.
* Evidence of skin conditions other than psoriasis (e.g., eczema) that could interfere with psoriasis assessments.
* History of chronic infection or malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Axis Clinical Trials, Los Angeles, California
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - The University of Utah, Salt Lake City, Utah
- Innovaderm Research Inc., Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Three patients in each of the 4 dose-escalating cohorts were randomized to receive placebo tablets that matched the active product in size and number (one 10 mg tablet, three 10 mg tablets, one 50 mg plus one 10 mg tablet, or two 50 mg tablets, respectively), daily for 12 weeks. The data of all placebo recipients were pooled for analyses.
- Apo805K1 10 mg: Patients in this treatment group received a single 10 mg tablet of Apo805K1 daily for 12 weeks
- Apo805K1 30 mg: Patients in this treatment group received three 10 mg tablets of Apo805K1 daily for 12 weeks
- Apo805K1 60 mg: Patients in this treatment group received one 10 mg tablet plus one 50 mg tablet of Apo805K1 daily for 12 weeks
- Apo805K1 100 mg: Patients in this treatment group received two 50 mg tablets of Apo805K1 daily for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Started | 12 | 12 | 12 | 12 | 12
Completed | 10 | 12 | 11 | 8 | 10
Not Completed | 2 | 0 | 1 | 4 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 1 | 1
Not completed — Sponsor concern over ECG result | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total of 60 patients were enrolled. No formal sample size calculation for this study was done, as this study was an exploratory study with main objective to assess the safety and tolerability of Apo805K1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 12 | 12 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8 | 3 | 0 | 19
  Male | 9 | 7 | 4 | 9 | 12 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 0 | 1 | 3 | 10
  White | 9 | 8 | 10 | 10 | 9 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 12 | 9 | 7 | 51
  Canada | 1 | 0 | 0 | 3 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Description: The number of patients in each treatment group who reported at least 1 adverse event, including clinically significant changes from baseline in vital signs, 12-lead ECG, physical examinations and laboratory tests, from the time of the first dose until the last study visit.
Time Frame: 12 Weeks
Population: The Safety Population consisted of all patients who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
participants | 4 | 5 | 7 | 6 | 5

2. Secondary Outcome: Cmax of Apo805K1 Following Multiple Doses, Assessed at Day 14
Description: Cmax for dosages of 10 mg, 30 mg, 60 mg, or 100 mg Apo805K1, determined on Day 14. Serial blood samples for PK analysis were collected pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose.
  .
Time Frame: 12 hours
Population: The Pharmacokinetics Population consisted of all patients who received Apo805K1 and provided evaluable PK data on at least one visit (Day 1 or Day 14)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/mL | 18.3 (9.7) | 53.0 (37.8) | 138.5 (54.5) | 164.9 (69.2)

3. Secondary Outcome: Tmax of Apo805K1 Following Multiple Doses, Assessed at Day 14
Description: Tmax for dosages of 10 mg, 30 mg, 60 mg, or 100 mg Apo805K1, determined on Day 14. Serial blood samples for PK analysis were collected pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose.
Time Frame: 12 hours
Measure: Median (Full Range); unit: hour
Arm/Group | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
hour | 4.00 [3.00 to 6.00] | 3.00 [3.00 to 5.00] | 3.00 [3.00 to 6.00] | 4.00 [3.00 to 6.00]

4. Secondary Outcome: AUC 0-infinity of Apo805K1 Following Multiple Doses, Assessed at Day 14
Description: AUC 0-infinity for dosages of 10 mg, 30 mg, 60 mg, or 100 mg Apo805K1, determined on Day 14. Serial blood samples for PK analysis were collected pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose.
Time Frame: 12 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng *hr/mL
Arm/Group | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 12
ng *hr/mL | 134.7 (68.1) | 368.4 (244.6) | 973.7 (463.1) | 1294.0 (658.7)

5. Secondary Outcome: T 1/2 of Apo805K1 Following Multiple Doses, Assessed at Day 14
Description: T 1/2 for dosages of 10 mg, 30 mg, 60 mg, or 100 mg Apo805K1, determined on Day 14. Serial blood samples for PK analysis were collected pre-dose and at 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose.
Time Frame: 12 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 12
hour | 2.8 (0.5) | 2.6 (0.2) | 2.8 (1.1) | 2.8 (0.5)

6. Secondary Outcome: Efficacy of Apo805K1 as Assessed by Change From Baseline in Psoriasis Area Severity Index (PASI) Scores
Description: PASI is a quantitative measure of psoriasis that combines an assessment of the severity of lesions and a measurement of how much of the body surface area is affected into a single score ranging from 0 (no disease) to 72 (maximal disease). Thus, a decrease in PASI score indicates improvement. This outcome measure compared the difference in change in PASI score from baseline to Week 12 between the active treatment groups and the placebo group.
Time Frame: Baseline to 12 Weeks
Population: The Efficacy Population was defined as all patients who received at least 1 dose of study medication and completed at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Three patients in each of the 4 dose-escalating cohorts were randomized to take placebo tablets that matched the active product in size and number (one 10 mg tablet, three 10 mg tablets, one 50 mg plus one 10 mg tablet, or two 50 mg tablets, respectively), daily for 12 weeks. The data of all placebo recipients were pooled for analyses.
- Apo805K1 10 mg: Patients in this treatment group took a single 10 mg tablet of Apo805K1 daily for 12 weeks
- Apo805K1 30 mg: Patients in this treatment group took three 10 mg tablets of Apo805K1 daily for 12 weeks
- Apo805K1 60 mg: Patients in this treatment group took one 10 mg tablet plus one 50 mg tablet of Apo805K1 daily for 12 weeks
- Apo805K1 100 mg: Patients in this treatment group took two 50 mg tablets of Apo805K1 daily for 12 weeks
Arm/Group | Placebo | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 12
units on a scale | -3.8 (4.6) | -3.8 (6.9) | -2.0 (5.3) | -3.4 (3.5) | -2.8 (5.0)
Statistical Analysis 1: Comparison: Placebo vs Apo805K1 10 mg vs Apo805K1 30 mg vs Apo805K1 60 mg vs Apo805K1 100 mg; The difference in change in PASI score from baseline to Week 12 was compared all active treatment groups and the placebo group; Test type: Superiority or Other; p = 0.9048, ANOVA

7. Secondary Outcome: Efficacy of APO805K1 as Assessed by Achievement of PASI-75
Description: The proportion of patients in each treatment group who achieved at least a 75% improvement in PASI score from baseline at Week 12
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 12
percentage of patients | 16.7 | 16.7 | 0.0 | 0.0 | 8.3
Statistical Analysis 1: Comparison: Placebo vs Apo805K1 10 mg vs Apo805K1 30 mg vs Apo805K1 60 mg vs Apo805K1 100 mg; Test type: Superiority or Other; p = 0.1975, Cochran-Armitage trend test

8. Secondary Outcome: Efficacy of Apo805K1 as Assessed by Change From Baseline at Week 12 in Lattice System-Physician Global Assessment (LS-PGA) Scores
Description: The LS-PGA is a standardized method for determining categories of psoriasis severity. The percentage of body surface area involved is assessed on a scale ranging from 1 (0%) to 7 (51-100%); measures of plaque severity (thickness, erythema, and scaling) are assessed using a 4-point scale ranging from "none" to "marked"; and an algorithm is used to combine the above scores to determine a final score on a scale ranging from 0 (clear) to 7 (very severe). Thus, a decrease in LS-PGA score indicates improvement. This outcome measure compared the difference in change in LS-PGA score from baseline to Week 12 between the active treatment groups and the placebo group.
Time Frame: Baseline to 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 12
units on a scale | -0.8 (0.8) | -1.2 (1.6) | -0.6 (0.7) | -0.5 (0.9) | -0.7 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Apo805K1 10 mg vs Apo805K1 30 mg vs Apo805K1 60 mg vs Apo805K1 100 mg; Test type: Superiority or Other; p = 0.6349, Kruskal-Wallis

9. Secondary Outcome: Efficacy of Apo805K1 as Assessed by Change From Baseline to Week 12 in Physician Global Assessment (PGA) Score
Description: In the PGA, the physician assigns a single estimate of a patient's overall severity of the disease using a scale ranging from 0 (Clear) to 7 (Severe). (Unlike the LS-PGA, the individual elements of psoriasis plaque morphology or degree of body surface area involvement are not quantified.) Thus, a decrease in PGA score indicates improvement. This outcome measure compared the difference in change in PGA score from baseline to Week 12 between the active treatment groups and the placebo group.
Time Frame: Baseline to 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 12
units on a scale | -1.0 (1.0) | -0.8 (1.0) | -0.5 (1.1) | -0.9 (0.8) | -1.3 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Apo805K1 10 mg vs Apo805K1 60 mg vs Apo805K1 100 mg; Test type: Superiority or Other; p = 0.6212, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected from the time of the first dose until the last study visit (Day 84) or following early withdrawal. Serious adverse events were collected up to 30 days after the last dose of study drug
Description: Patients were provided with a diary card in which to record AEs, and were questioned at each visit. Vital signs, ECG, physical examination findings, and laboratory parameters were assessed for changes from baseline of clinical significance.
Arm/Group | Placebo | Apo805K1 10 mg | Apo805K1 30 mg | Apo805K1 60 mg | Apo805K1 100 mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 1/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 5/12 | 7/12 | 6/12 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Apo805K1 10 mg (N=12) | Apo805K1 30 mg (N=12) | Apo805K1 60 mg (N=12) | Apo805K1 100 mg (N=12)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Apo805K1 10 mg (N=12) | Apo805K1 30 mg (N=12) | Apo805K1 60 mg (N=12) | Apo805K1 100 mg (N=12)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic nerve cupping (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days